CLINICAL TRIAL: NCT06822725
Title: The Sinonasal Microbiome
Status: Active, not recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 09-354-A
Record Dates: First submitted 2025-01-28; First posted 2025-02-12 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Sinonasal Disorder; Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease | interventions — Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic rhinosinusitis (CRS) with and without Nasal Polyposis: Those with and without nasal polyps, and those with acute exacerbations
  Interventions: Procedure: Chronic rhinosinusitis (CRS) with and without Nasal Polyposis
- Control Group: Normals without allergy, those with perennial allergic rhinitis
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Control Group — normals without allergy, those with perennial allergic rhinitis
  Groups: Control Group
Procedure: Chronic rhinosinusitis (CRS) with and without Nasal Polyposis — Those with and without nasal polyps, and those with acute exacerbations
  Groups: Chronic rhinosinusitis (CRS) with and without Nasal Polyposis

SUMMARY:
Chronic rhinosinusitis is an inflammatory disease of the sinonasal mucosa with significant impact and limited treatment options. Chronic rhinosinusitis (CRS) poses an important public health problem and causes a large impact on individual quality of life. Studies of CRS have been limited by access to tissue, the complexity of the sinonasal physiology, a lack of available biomarkers, the absence of useful animal models, a paucity of cohorts with biological samples for analysis, and limited well-designed clinical trials or investigations of immune function. Therefore, novel strategies for identifying biological mechanisms underlying this disease are in great need.

Using prospective samples from well characterized subjects, the investigators intend to profile the mucosa associated-bacteria in the nose and sinuses. In parallel, using sinus tissue from patients undergoing surgery, the site will interrogate the epithelium for mucosal immune function to understand host-microbe interaction. This study hypothesizes that the microbial profile of the sinuses initiates an immune responses which leads to chronic inflammation in susceptible people. This study would provide the first comprehensive data on what bacteria are present in the nose and sinus and could lead to important knowledge useful in sinonasal disease.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Diagnosis of chronic sinusitis (with or without nasal polyposis), perennial allergic rhinitis, or normal sinuses/absence of allergy

Exclusion Criteria:

* Use of immunosuppressants
* Immunodeficiency
* Inability to stop sinusitis related medications for 10 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will examine the sinonasal microbiota in subjects with CRS (at baseline in those with and without nasal polyps, and those with acute exacerbations) and controls (normals without allergy, those with perennial allergic rhinitis).
Sampling Method: Probability Sample
Enrollment: 285 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Determining the distinct bacterial profiles with abundance of organisms using the Pyrosequencing Pipeline service | At baseline until final values at 36 months.
Determining the distinct bacterial profiles with shift toward anaerobic bacteria using the Pyrosequencing Pipeline service | At baseline until final values at 36 months.
Determining the distinct bacterial profiles with lower bacterial diversity using the Pyrosequencing Pipeline service | At baseline until final values at 36 months.

SECONDARY OUTCOMES:
the discovery of low frequency and novel organisms using the Pyrosequencing Pipeline service | At baseline until final values at 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jayat Pinto, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Hyde Park, Illinois, United States